CLINICAL TRIAL: NCT04213157
Title: Evaluation Trifecta and Pentafecta Outcomes of Patients Underwent Laparoscopic Partial Nephrectomy for cT1 Renal Tumor
Brief Title: Laparoscopic Partial Nephrectomy for cT1 Tumors
Status: Completed | Type: Observational
Sponsor: Samsun Liv Hospital (Other)
Collaborators: Ondokuz Mayıs University (Other)
Responsible Party: Principal Investigator, Mehmet Necmettin Mercimek, Principal Investigator, Samsun Liv Hospital
Other Study IDs: OMU KAEK 2019/241
Record Dates: First submitted 2019-12-25; First posted 2019-12-30 (Actual); Last update posted 2020-01-02 (Actual); Status verified 2019-12

CONDITIONS: Renal Cancer; Renal Neoplasm; Renal Cell Carcinoma; Surgery; Surgery--Complications; Renal Functional Abnormality; Oncology; Oncology Problem; Kidney Ischemia; Kidney Injury; Urologic Neoplasms; Urologic Cancer; Kidney Neoplasms
Keywords: laparoscopic partial nephrectomy; Trifecta; Pentafecta; Outcomes
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell; Neoplasms; Urologic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aim of the study is to evaluate trifecta and pentafecta outcomes for laparoscopic partial nephrectomy (LNP) in patients with clinical T1N0M0 renal tumor.

DETAILED DESCRIPTION:
From November 2009 to August 2018 a total of 292 patients who underwent LPN by global ischemia were included in the study. The patients were allocated into two groups according to the tumor size; T1a (≤ 40 mm, n=215), T1b (41-70 mm, n=77). Demographics features, clinical tumor characteristics, intraoperative and postoperative outcomes were analyzed. A negative surgical margin, warm ischemia time (WIT) < 20 min and no postoperative complications (Clavien-Dindo ≥ grade 3) were accepted to achieve the trifecta outcomes. Pentafecta has defined as trifecta criteria plus >90% preservation of estimated glomerular filtration rate (eGFR) and no stage upgrade of chronic kidney disease 12 months after LPN. Univariable and multivariable analysis were used to identify factors predicting trifecta and pentafecta achievement.

ELIGIBILITY:
Inclusion Criteria:

* Functioning contraleteral kidney
* Patients with complete data
* Patients with single renal tumor on the effected side
* Patients who approved the written consent form

Exclusion Criteria:

* The patients with bilateral renal tumors (n=8, 16 LPNs)
* solitary kidney (n=8)
* horseshoe kidney (n=4)
* pelvic ectopic kidney (n=2)
* graft kidney (n=2)
* those with multiple renal tumors in a single kidney (n=3) or with > 7 cm renal tumor (n=6)
* Patients who were operated on for colon cancer (n=4), prostate cancer (n=2), endometrial cancer (n=1) or adrenal mass (n=2) within the first year after LPN

Ages: 18 Years to 82 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Two hundred ninety-two patients who have a follow-up at least 12 months were included in the study. Those were allocated into two groups according to radiological tumor size; 215 patients with tumor size ≤ 40 mm were included in group T1a and 77 patients with tumor size 41-70 mm were included in group T1b.
Sampling Method: Probability Sample
Enrollment: 292 (Actual)
Dates: Start 2019-03-15 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2019-11-10 (Actual)

PRIMARY OUTCOMES:
Operation time | at the end of the surgery
  time from onset to complete of surgery
Blood loss | at the end of the surgery
  amount of bleeding during surgery (mL)
warm ischemia time | at the and of the surgery
  The clamp time of the renal artery and vein which is required to complete tumor excision and renorrhaphy
intraoperative complication | at the end of the surgery
  abnormal problmes that may be seen during surgery
Postoperative complication | up to 3 months
  abnormal problmes that may be seen after surgery and require additional intervention, treatment or follow-up
functional outcomes | up to 1 year postoperatively
  serum creatinine level and estimated glomerular filtration rate
surigcal margin status | up to 1 month postoperatively
  presence or absence of tumors at the surgical margin
Relative decrease in renal function | up to 1 year postoperatively
  Comparison of preoperative and postoperative renal functions according to numerical and percentile values
CKD stage upgrading | up to 1 year postoperatively
  evaluation of preoperative and postoperative renal functions according to chronic kidney disease stages
Oncological outomes | up to the last clinical control (months)
  Presence or absence of local and/or distal tumor recurrence

CONTACTS AND LOCATIONS:
Overall Officials: Saban Sarıkaya, Professor, Study Chair — Ondokuz Mayıs University; Ender Ozden, Professor, Study Director — Ondokuz Mayıs University
Locations (2):
- Turkey (Türkiye) (2):
  - Liv hospital samsun, Samsun
  - Ondokuz Mayıs University, Samsun

IPD SHARING:
Plan to Share IPD: Undecided
It is not yet known if there will be a plan to make IPD available.

REFERENCES:
- [Result] Porpiglia F, Bertolo R, Amparore D, Fiori C. Margins, ischaemia and complications rate after laparoscopic partial nephrectomy: impact of learning curve and tumour anatomical characteristics. BJU Int. 2013 Dec;112(8):1125-32. doi: 10.1111/bju.12317. Epub 2013 Aug 13. PMID 23937616
- [Result] Minervini A, Siena G, Antonelli A, Bianchi G, Bocciardi AM, Cosciani Cunico S, Ficarra V, Fiori C, Fusco F, Mari A, Martorana G, Medica M, Mirone V, Morgia G, Porpiglia F, Rocco F, Rovereto B, Schiavina R, Simeone C, Terrone C, Volpe A, Carini M, Serni S; Members of the RECORd Project-LUNA Foundation. Open versus laparoscopic partial nephrectomy for clinical T1a renal masses: a matched-pair comparison of 280 patients with TRIFECTA outcomes (RECORd Project). World J Urol. 2014 Feb;32(1):257-63. doi: 10.1007/s00345-013-1155-7. Epub 2013 Sep 7. PMID 24013181
- [Result] Osaka K, Makiyama K, Nakaigawa N, Yao M. Predictors of trifecta outcomes in laparoscopic partial nephrectomy for clinical T1a renal masses. Int J Urol. 2015 Nov;22(11):1000-5. doi: 10.1111/iju.12893. Epub 2015 Aug 6. PMID 26251228
- [Result] Rais-Bahrami S, Romero FR, Lima GC, Kohanim S, Permpongkosol S, Trock BJ, Jarrett TW, Kavoussi LR. Elective laparoscopic partial nephrectomy in patients with tumors >4 cm. Urology. 2008 Sep;72(3):580-3. doi: 10.1016/j.urology.2008.05.027. Epub 2008 Jul 16. PMID 18632142
- [Derived] Mercimek MN, Ozden E, Gulsen M, Yakupoglu YK, Bostanci Y, Sarikaya S. Which Is the Best Predictor to Achieve Trifecta in Patients Undergoing Elective Laparoscopic Partial Nephrectomy with Global Hilar Clamping? Comparative Analysis in Patients with Clinical T1a and T1b Renal Tumors. J Endourol. 2021 May;35(5):615-622. doi: 10.1089/end.2020.0758. Epub 2020 Nov 5. PMID 32967451